CLINICAL TRIAL: NCT02236663
Title: Effectiveness of a Safety App to Respond to Dating Violence for College Women and Their Friends
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Arizona State University (Other); University of Missouri-Columbia (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NA_00054334; 1R01HD076881-01A1 (NIH)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Intimate Partner Violence
Keywords: Intimate Partner Violence; Dating Violence; Relationships; Safety Planning; College; Student; App
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- App Based Safety Decision Aid (Experimental): Personalized App-Based Safety Decision Aid
  Interventions: Behavioral: Personalized App-Based Safety Decision Aid
- Control App (Active Comparator): Usual Care Safety Plan
  Interventions: Behavioral: Usual Care Safety Planing App

INTERVENTIONS:
Behavioral: Usual Care Safety Planing App — The control group App will provide women and friends with basic safety planning information and a brief resource list of IPV resources. The resources will be targeted to college students age 18-24 years. The control group App safety plan is not personalized to woman/friend's safety priorities and danger in the relationship.
  Arms: Control App
Behavioral: Personalized App-Based Safety Decision Aid — Setting of priorities for safety: participants will establish priorities by making pairwise comparisons of importance between 5 factors.
  Danger Assessment: asks participants to report on well-established risk factors for repeat violence and lethal IPV. A weighted scoring algorithm provides participants with their validated level of danger and safety planning information and resources based on their level of danger.
  Personalized action plan: Based on a participant's answers to the previous sections, a list of safety strategies with links to resources will be presented tailored to their level of danger and priority settings. The participant is given the option to print results and the personalized plan.
  Arms: App Based Safety Decision Aid

SUMMARY:
Intimate partner violence (IPV), including violence in dating relationships (dating violence, DV) is a widespread and serious public health problem. Among U.S. female IPV survivors, 47.1% report their first abusive relationship occurred at college age (age 18-24). Similarly, in national surveys, adults respondents 18-24 years of age report the highest rate of stalking victimization, most commonly by a former intimate partner. Safety planning is the most widely used intervention to prevent and respond to IPV, yet the vast majority of abused women never access safety planning services. Our challenge is to increase college women's access to safety planning, with the opportunity to consider their unique safety priorities and level of danger during and when ending an abusive relationship. In addition, while "bystander" interventions that train peers to safely intervene have been shown to be effective in sexual assault prevention on campus, and college women in abusive relationships most frequently disclose IPV to a friend, no similar interventions have been tested with friends for IPV response on campuses. Therefore, the objective of the study is to evaluate the:

1. effectiveness of an interactive, personalized smart phone and web based safety application ("App") intervention in Maryland and Oregon with: 1) college women (age 18-24) who experience IPV and 2) friends (age 18-24) of women experiencing IPV. The safety decision App allows the user to enter information on: a) relationship health; b) safety priorities; and c) severity of violence/danger in relationship. The App then uses the information to provide the user with a personalized safety planning information and resources; and
2. dissemination of the App nationally to determine the reach, adoption, implementation and maintenance of App use among university/college students.

ELIGIBILITY:
Inclusion Criteria:

* Females who report current physical violence, sexual violence, psychological abuse or stalking by a dating/intimate/ex-intimate partner, or who have a female friend currently experiencing abuse from dating/intimate/ex-intimate partner.
* Males who have a female friend currently experiencing physical violence, sexual violence, psychological abuse or stalking by a dating/intimate/ex-intimate partner
* English speaking
* Between the ages of 18-24 years old
* Attend a college in Maryland or Oregon
* Enrolled in college or university (at least part time)
* Have access to a safe smart-phone or computer with internet and are comfortable downloading an app or using the internet
* Have a safe email address

Exclusion Criteria:

* Younger than 18 years of age
* Older than 24 years of age
* Cannot read/speak English
* Live outside targeted states
* No access to safe smart phone or computer with internet
* Uncomfortable with downloading an app
* No access to a safe email address
* Does not report current violence from an intimate partner or having a female friend that has experienced intimate partner violence

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 649 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in survivors' use of safety strategies on Safety Behavior Checklist at 12 months | Baseline, 12 Months
  Adapted from Intimate Partner Violence Strategies Index to assess for survivors the range of strategies used to halt, escape, or resist violence, and the helpfulness of each strategy.
Change from baseline in survivors' and friends' decisional conflict on Decisional Conflict Scale (DCS) immediately post intervention. | Baseline, immediately post intervention
  The DCS consists of twelve items, with each question having three response options (yes, no, and unsure). The DCS provides a total score, which is a measure of the decision process, as well as scores for four subscales (feeling informed, certainty about decision, values clarity, and support), with higher scores on the DCS indicating a greater degree of decisional conflict (indicative of a poorer decision process). Will be used to assess decisional conflict with survivors and friends.
Change from baseline in friends' efficacy to intervene on adapted Self-efficacy to Deal with Violence Scale at 12 months | Baseline, 12 months
  19 times scale adapted to assess friends of survivors' confidence to intervene.
Changes from baseline in friends' supportive behaviors on Supportive Behaviors Checklist at 12 months | Baseline, 12 months
  Assesses supportive behaviors used to assist a friend experiencing intimate partner violence.

SECONDARY OUTCOMES:
Change from baseline in survivors' drug and alcohol use on adapted Monitoring the Future Drug and Alcohol Questionnaire at 12 months. | Baseline, 12 months
Change from baseline in survivors' abuse exposure on the Composite Abuse Scale (CAS) at 12 months | Baseline, 12 months
  The CAS is a 30 item validated comprehensive intimate partner violence screening measure with
Change from baseline in survivors' and friends' Decisional Conflict on Decisional Conflict Scale at 12 mo | Baseline, 12 month
Change from baseline in survivor' depression on Center for Epidemiologic Studies Depression Scale, Revised at 12 months | Baseline, 12 months
  A 20-item self report measure, designed to screen for depressive symptoms in community samples and assess the probability that an individual meets the criteria for major depressive disorder.
Changes from baseline in friends' attitudes on the Intimate Partner Violence on the Acceptance of Dating Violence Scale at 12 months | Baseline, 12 months
  5 item scale used to measures norms that support violence.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Glass, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (4):
- United States (4):
  - Arizona State University, Phoenix, Arizona
  - Johns Hopkins University School of Nursing, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Kaiser Foundation Research Institute, Portland, Oregon

REFERENCES:
- [Derived] Bloom TL, Perrin N, Brown ML, Campbell J, Clough A, Grace KT, Laughon K, Messing J, Eden KB, Turner R, Glass N. Concerned friends of intimate partner violence survivors: results from the myPlan randomized controlled trial on college campuses. BMC Public Health. 2023 May 31;23(1):1033. doi: 10.1186/s12889-023-15918-y. PMID 37259087
- [Derived] Glass NE, Clough A, Messing JT, Bloom T, Brown ML, Eden KB, Campbell JC, Gielen A, Laughon K, Grace KT, Turner RM, Alvarez C, Case J, Barnes-Hoyt J, Alhusen J, Hanson GC, Perrin NA. Longitudinal Impact of the myPlan App on Health and Safety Among College Women Experiencing Partner Violence. J Interpers Violence. 2022 Jul;37(13-14):NP11436-NP11459. doi: 10.1177/0886260521991880. Epub 2021 Feb 12. PMID 33576291
- [Derived] Glass N, Clough A, Case J, Hanson G, Barnes-Hoyt J, Waterbury A, Alhusen J, Ehrensaft M, Grace KT, Perrin N. A safety app to respond to dating violence for college women and their friends: the MyPlan study randomized controlled trial protocol. BMC Public Health. 2015 Sep 8;15:871. doi: 10.1186/s12889-015-2191-6. PMID 26350482